CLINICAL TRIAL: NCT06388421
Title: DeciPHer-ILD: A Real-world Patient Registry in Group 3 Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Status: Recruiting | Type: Observational
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: GMS-PH-401
Record Dates: First submitted 2024-04-12; First posted 2024-04-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension Due to Lung Diseases and Hypoxia; Pulmonary Hypertension; Interstitial Lung Disease
Keywords: pulmonary hypertension; interstitial lung disease; pulmonary hypertension associated with interstitial lung disease
MeSH Terms: conditions — Hypoxia; Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For patients consenting to genomic analysis, a blood sample will be collected. These samples will be shipped to the central laboratory for processing and storage prior to analysis. Genomic analysis will be analyzed for genetic markers that may be associated with clinical response and tolerability.
  For patients consenting to optional biomarker sample, blood will be collected for the evaluation of biomarkers (specific targets to be determined).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Cohort 1: Cohort 1 will include approximately 500 patients who are not receiving inhaled treprostinil at time of study enrollment.
  Interventions: Other: Prospective study assessments
- Cohort 2: Cohort 2 will include approximately 150 patients who are newly initiated on Tyvaso/Tyvaso DPI. For patients to be eligible for Cohort 2, they must have initiated Tyvaso/Tyvaso DPI at Baseline or ≤ 60 days prior to Baseline.
  Interventions: Other: Prospective study assessments
- Cohort 3: Cohort 3 will include approximately 350 patients who have been receiving Tyvaso/Tyvaso DPI for > 60 days prior to Baseline.
  Interventions: Other: Prospective study assessments

INTERVENTIONS:
Other: Prospective study assessments — Patients will complete prospective assessments at 6- and 12-month intervals for up to 5 years. There will be 1 check in at the first 3 months of enrollment. Follow up visits will include a ±45 day visit window. If an assessment is performed within 45 days of the visit window as part of the patient's standard of care, those values will be used in place of a prospective assessment.

SUMMARY:
This is a prospective, non-interventional, multicenter, registry of patients with pulmonary hypertension associated with interstitial lung disease (PH-ILD).

DETAILED DESCRIPTION:
The purpose of this study is to observe and capture demographic characteristics, treatment patterns, and clinical outcomes of interest for patients with PH-ILD to further clinical understanding of the epidemiological landscape and outcomes of the disease and treatment.

In this registry, patients will be enrolled into 1 of 3 cohorts. Cohort 1 will include approximately 500 patients who are not receiving inhaled treprostinil at time of study enrollment. Cohort 2 will include approximately 150 patients who are newly initiated on Tyvaso/Tyvaso DPI. Cohort 3 will include approximately 350 patients who have been receiving Tyvaso/Tyvaso DPI for >60 days.

As part of the registry, assessments will be completed for data collection in 6- or 12 month intervals, unless the data are already available via standard of care. This patient registry will follow patients for up to 5 years after enrollment.

Assessments include pulmonary function tests (PFTs) including diffusing capacity of the lungs for carbon monoxide (DLCO); high resolution computed tomography (HRCT); vital signs; 6-Minute Walk Test; blood draw for plasma N-terminal pro-BNP (NT-proBNP) concentration, genetics analysis, biomarker analysis; echocardiography; EuroQoL 5 Dimension 5 Level Questionnaire (EQ-5D-5L); King's Brief Interstitial Lung Disease Questionnaire (K-BILD); Living with Pulmonary Fibrosis Questionnaire (L-PF); Therapy Administration Questionnaire; healthcare resource utilization; current medications and rehabilitation; WHO functional class; transplant status; survival data; and RHC.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Diagnosis of ILD by traditional or HRCT determined by the site/institution that conducted the HRCT
3. Patients with connective tissue disease must have a baseline forced vital capacity of <70%
4. RHC confirmed PH (mean pulmonary artery pressure >20 mmHg, pulmonary arterial wedge pressure ≤15 mmHg, pulmonary vascular resistance >2 WU).
5. For patients to be eligible for Cohort 1, they must not be receiving inhaled treprostinil at Baseline.
6. For patients to be eligible for Cohort 2, they must have initiated Tyvaso/Tyvaso DPI at 1 of the following time points:

   1. Baseline
   2. ≤60 days prior to Baseline
7. For patients to be eligible for Cohort 3, they must be receiving Tyvaso/Tyvaso DPI at Baseline and for >60 days prior to Baseline
8. Co-enrollment in other observational or interventional studies is permitted
9. Patient is willing and able to provide informed consent and complete surveys/questionnaires in English or Spanish

Exclusion Criteria:

1. Confirmed diagnosis of Group 1, 2, 4, or 5 PH
2. Confirmed diagnosis of Group 3 PH related to chronic obstructive pulmonary disease or conditions that cause hypoxemia, such as untreated or inadequately treated obstructive sleep apnea and alveolar hypoventilation disorders
3. Patients receiving Yutrepia (inhaled treprostinil) at Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of pulmonary hypertension associated with interstitial lung disease. This includes patients who are and aren't receiving inhaled treprostinil, excluding patients receiving Yutrepia™ at Baseline.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristics as described by demographics, medical history, ILD history, PH history, family history (comorbidities), and diagnostic right heart catheterization values | Baseline

SECONDARY OUTCOMES:
Changes in clinical features relating to patients' interstitial lung disease and pulmonary hypertension | Followed prospectively for a maximum of 5 years from date of enrollment into the registry

CONTACTS AND LOCATIONS:
Locations (59):
- United States (58):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Health - University Medical Center Phoenix, Phoenix, Arizona
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - NCH Research Institute, Naples, Florida
  - Advent Health Medical Group Advanced Lung Disease, Orlando, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Tampa General Hospital/University of South Florida Health, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University Medical Center - New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Northwell Health, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Pulmonix, LLC, Greensboro, North Carolina
  - East Carolina University Health, Greenville, North Carolina
  - Wakemed Health and Hospital, Raleigh, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Ohio State Richard M. Ross Heart Hospital, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Summit Health, Bend, Oregon
  - Legacy Research Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Sidney Kimmel Medical College, Philadelphia, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - StatCare Pulmonary Consultants and Center for Biomedical Research, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwest Medical Center Heart and Lung Clinic, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Inova Medical Group, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Marshall Health, Huntington, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Auxilio Mutuo Hospital, Guaynabo, Puerto Rico, Puerto Rico